CLINICAL TRIAL: NCT01226407
Title: Phase I Study of CG200745 to Examine the Maximum Tolerate Dose, Pharmacokinetic and Pharmacodynamic Profiles, and Safety Among Patients With Progressive Solid Cancer
Brief Title: Examine Maximum Tolerated Dose and Pharmacokinetic and Pharmacodynamic Profile
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG200745-1-01
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-10

CONDITIONS: Solid Tumour
Keywords: Solid Tumour
MeSH Terms: interventions — N1-(3-(dimethylamino)propyl)-N8-hydroxy-2-((naphthalene-1-loxy)methyl)oct-2-enediamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm for CG200745 (Experimental): any progrossive solid cancer
  Interventions: Drug: CG200745

INTERVENTIONS:
Drug: CG200745 — Multiple administration (IV) over the cycles untile MTD/LTD
  Other Names: No specific generic name yet

SUMMARY:
Open label, single dose and phase I study.

The primary objective: To determine the maximum tolerated dose in Single dose

The secondary objective: to evaluate the toxicity in administration to determine desirable dosing amount for phase II to evaluate tumor response in progressive solid cancer patients to evaluate pharmacokinetic/ pharmacodynamic profile.

DETAILED DESCRIPTION:
1. Number of Subjects: 28~36, dose escalation (2~6 subject of each step)
2. Adverse Events will be coded to preferred therm and body system using the CTCAE

ELIGIBILITY:
Inclusion Criteria:

* from 20 years old to 69 years old
* diagnosed with progressive solid cancer
* In spite of standard chemotherapies, the efficacy of the treatment or life extension cannot be expected.
* Evaluated 0-1 of ECOG
* Expected life duration is within 3 months

Exclusion Criteria:

* Major surgery except tumor-removal surgery received within 2 weeks of screening.
* history of CNS metasis
* hyper-sensitivy of study drug
* pregancy or lactating
* administered other HDAC inhibitor within 4 weeks of screening

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose in Single dose | On 22 days after administration

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, MD, PhD, Principal Investigator — Seoul Asan medical Center
Locations (1):
- Seoul Asan Medical Center, Seoul, South Korea